CLINICAL TRIAL: NCT05271877
Title: Evaluation of Surgical and Obstetric Outcomes in Pregnant Women Undergoing Operative Laparoscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, M.D. Ph.D., Università degli Studi dell'Insubria
Other Study IDs: LAPRE-1
Record Dates: First submitted 2022-02-27; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Pregnancy Related; Laparoscopy
Keywords: Pregnancy; Laparoscopy
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women, regardless of the gestational age.
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Laparoscopy — Diagnostic/operative laparoscopic procedure

SUMMARY:
Laparoscopy, when applicable, is the current gold standard management for abdominal and pelvic surgery. Although accumulating evidence suggests that laparoscopy is associated with reduced intraoperative and postoperative morbidity, reduced hospital stay, better recovery and cosmesis compared with open surgery (laparotomy), the use of this technique in pregnant women is still debated. Considering this point, we aimed to collect retrospectively cases of laparoscopic surgery during pregnancy, regardless of the indication and gestational age, in order to analyze both surgical and obstetric outcomes during and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (regardless of gestational age)
* At least one indication for laparoscopic surgery

Exclusion Criteria:

* None

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women undergoing laparoscopy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Intraoperative complication | From the beginning to the end of laparoscopy
  Any complication during laparoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Ph.D., Principal Investigator — Università degli Studi dell'Insubria

IPD SHARING:
Plan to Share IPD: Undecided